CLINICAL TRIAL: NCT04035382
Title: BMI-Associated Labor Induction: A Prospective Trial
Acronym: BALI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baystate Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BH-19-000
Record Dates: First submitted 2019-07-16; First posted 2019-07-29 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Labor Induction
Keywords: BMI; Obesity; Labor induction; Cesarean section
MeSH Terms: conditions — Obesity | interventions — Labor, Induced; Misoprostol; Oxytocin; Amniotomy

STUDY DESIGN:
Intervention Model Description: Simon two-stage
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Labor Induction (Experimental): Induction of labor between 39 0/7 to 39 6/7 weeks. Cervical ripening and induction method will be left to the managing clinician. However, combination method of cervical ripening with prostaglandin or oxytocin and Foley catheter, followed by oxytocin infusion and amniotomy will be encouraged.
  Interventions: Procedure: Labor induction

INTERVENTIONS:
Procedure: Labor induction — The study intervention is labor induction from 39 0/7 to 39 6/7 weeks. The individual labor induction process will be at the discretion of the physician or midwife managing the subject's care. Methods of induction that may be used include misoprostol, intracervical Foley catheter, oxytocin, and/or amniotomy. Participating clinicians will be encouraged to use only one course of cervical ripening followed by oxytocin infusion and amniotomy.
  Other Names: Foley catheter; Misoprostol; Oxytocin; Amniotomy

SUMMARY:
The primary objective of this study is to determine if planned induction of labor at 39 weeks for nulliparous with pre-pregnancy BMI ≥ 35 kg/m2 reduces the incidence of cesarean section compared to expectant management

DETAILED DESCRIPTION:
Obesity in the obstetric population has reached epidemic proportions, affecting over 30% of reproductive-aged women in the United States (1). The increase in this morbidity is associated with large increases in cesarean delivery over the non-obese obstetric population and resultant post-operative complications are also higher in obese women (2). There are no interventions proven to reduce the risk of cesarean in obese women. The aim of this research study is to determine if induction of labor at 39 weeks can reduce the incidence of cesarean delivery over routine obstetric care (expectant management).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older
2. Pregnant, singleton gestation, vertex presentation
3. Nulliparous (no prior pregnancy delivered past 20 weeks)
4. Pre-pregnancy (self-reported in record of in EMR within 3 months of LMP) or 1st trimester (up to and including 14 weeks 0 days) BMI ≥ 35 kg/m2
5. Gestational age at enrollment 38 weeks 0 days and 38 weeks 6 days with dating confirmed by LMP and ultrasound performed prior to 20 6/7 weeks

Exclusion Criteria:

1. Plan for induction of labor prior to 41 weeks 0 days for medical indication prior to study consideration
2. Plan for cesarean delivery or contraindication to labor
3. Major illness with increased risk of adverse pregnancy outcomes (e.g. pregestational diabetes with or without medication, gestational diabetes on medication, hypertension, cardiac disease, renal insufficiency, autoimmune disorder)
4. Multiple gestation
5. Non-vertex presentation
6. Fetal death
7. Fetus with major/lethal anomaly or aneuploidy (soft markers of aneuploidy, urinary tract dilation, isolated bowel dilation, mild ventriculomegaly, normal variants of vascular system, and isolated ventricular septal defects will not be excluded)

   a. Soft markers not qualifying as exclusion criteria: echogenic intracardiac focus, choroid plexus cyst, echogenic bowel, increased NT or nuchal fold, isolate short humerus or femur
8. Fetal growth restriction (EFW <10th percentile or AC <10th percentile)
9. Preeclampsia or gestational hypertension
10. Known oligohydramnios or polyhydramnios
11. Prior delivery after 20 weeks
12. Placenta/vasa previa
13. Placental abruption (known or suspected) or unexplained vaginal bleeding
14. Previous cesarean section, myomectomy, or classical cesarean
15. Spontaneous labor or suspicion of labor with regular contractions and cervical change, rupture membranes
16. Active genital herpes or HIV positive
17. Inability to consent
18. Any contraindication to a vaginal delivery
19. Delivery anticipated outside of Baystate Medical Center

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2019-10-31 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of cesarean section | Admission for induction to discharge from delivery admission, up to 3 weeks after enrollment.
  The primary outcome is to determine whether planned induction of labor at 39 weeks for obese nulliparous women changes the incidence of cesarean section.

SECONDARY OUTCOMES:
Incisional extensions at cesarean section | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
  J or T shape incisions or cervical trauma
Operative vaginal delivery and indication | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
  Vacuum or forceps
Suspected intraamniotic infection | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
  At least one maternal fever ≥100.4 F with at least one additional clinical sign of maternal tachycardia, fetal tachycardia, uterine tenderness or purulent/foul smelling vaginal discharge
3rd or 4th degree perineal laceration | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Maternal death | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Antepartum, intrapartum, or neonatal death | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Admission to the intensive care unit (ICU) | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Preeclampsia | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
  Preeclampsia without severe features: Elevated blood pressure after 20 weeks ≥140/90 on 2 occasions at least 4 hours apart with previously normal blood pressure AND,
  * proteinuria (≥300 mg per 24 hours collection OR ≥0.3 mg/dL on protein:creatinine ratio OR 1+ on dipstick if neither of the previous is available)
  Preeclampsia with severe features: Elevated blood pressure after 20 weeks ≥160/110 on 2 occasions (may be within minutes to ensure medication treatment) OR,
  * Blood pressure ≥140/90 and systemic findings including: new platelet count <100,000microliter, serum creatinine >1.1 mg/dL, doubling of serum creatinine in absence of other renal disease, liver transaminases twice upper limit of normal, pulmonary edema, cerebral or visual symptoms
  * Proteinuria is not necessary for this diagnosis
  Eclampsia: preeclampsia with eclamptic seizure
Gestational hypertension | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
  Gestational hypertension: blood pressure elevation ≥140/90 on two occasions after 20 weeks in absence of proteinuria or systemic findings defined above
Postpartum hemorrhage | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
  Visual estimated blood loss >1000 mL or need for two or more uterotonics
Postpartum endometritis | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Composite maternal infectious outcome | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
  Endometritis, wound reopened for hematoma, seroma, infection, or other reasons, cellulitis requiring antibiotics, pneumonia, pyelonephritis, bacteremia of unknown source, septic pelvic thrombosis
Maternal venous thromboembolism | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Birth weight | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
  Macrosomia >4500 grams, large for gestational age (LGA) defined as 90th percentile weight for gestational age, assessed specifically by sex and race of the infant based on United States birth certificate data
Duration and presence (up to 72 hours) of respiratory support | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
  Including ventilator, CPAP, high-flow nasal cannula (HFNC)
Small for gestational age | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
  <5th percentile and <10th percentile weight for gestational age, assessed specifically by sex and race of the infant based on United States birth certificate data
Cephalohematoma | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Shoulder dystocia | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
  Need for additional maneuvers to accomplish delivery
Transfusion of blood products | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Breastfeeding intention and initiation in the hospital | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Breastfeeding at 6 weeks (exclusive and any breastfeeding) | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Hyperbilirubinemia requiring phototherapy or exchange transfusion | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Apgar ≤ 7 at 5 minutes | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Neonatal seizures | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Sepsis | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
  Requires the presence of a clinically ill infant in whom systemic infection is suspected with a positive blood, cerebrospinal fluid (CSF), or catheterized/suprapubic urine culture; or, in the absence of positive cultures, clinical evidence of cardiovascular collapse or an unequivocal X-ray confirming infection.
Neonatal encephalopathy | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
  As defined by Shankaran et al.
Meconium aspiration syndrome | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Birth trauma | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
  Bone fractures, brachial plexus palsy, other neurologic injury, retinal hemorrhage facial nerve injury
Intracranial hemorrhage or subgaleal hemorrhage | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Neonatal hypotension requiring pressor support | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Neonatal composite outcome | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
  IUFD, neonatal death, intubation or neonatal respiratory support, Apgar score ≤ 7 at 5 minutes, seizures, sepsis as defined above, neonatal encephalopathy, pneumonia, meconium aspiration syndrome, birth trauma, intracranial hemorrhage, or hypotension
Hypoglycemia | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
  glucose < 35 mg/dL requiring IV therapy
Admission to the neonatal intensive care unit (NICU) | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Number of clinic visits post enrollment to admission for delivery | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Non-stress tests, biophysical profiles (BPP), modified BPPs, ultrasounds done other than BPP, Doppler, contraction stress test | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Intrauterine pressure catheter (IUPC) or fetal scalp electrode placement | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Epidural use | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Use of induction and ripening agents, maximum dose of oxytocin | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Number of hours on labor and delivery unit | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Maternal postpartum length of hospital stay | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Neonatal length of hospital stay | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Length of NICU or intermediate care stay | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
Post discharge resource utilization | From enrollment to 6-8 weeks postpartum, average of 10 weeks after enrollment.
  Inpatient and outpatient visits for mother and baby from discharge to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Corina Schoen, MD, Principal Investigator — Baystate Medical Center
Locations (2):
- United States (2):
  - Baystate Medical Center, Springfield, Massachusetts
  - Sidney Kimmel Medical College, Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No